CLINICAL TRIAL: NCT00837135
Title: Pilot Study Of Safety And Feasibility Of GI-4000, An Inactivated Recombinant Saccharomyces Cerevisiae Expressing Mutant Ras Protein Combined With Adoptive Transfer And Chemoradiation in Locally Advanced Pancreatic Cancer
Brief Title: GI-4000 With Adoptive Transfer in Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to transfer of Investigator
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 806693; UPCC 03207
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- All Subjects (Experimental): Screening for Eligibility into Trial
  Interventions: Other: Screening
- ARM A (Experimental): GI-4000 Vaccine
  Interventions: Biological: GI-4000 Vaccine
- ARM B (Experimental): GI-4000 Vaccine + Activated T Cells
  Interventions: Biological: GI-4000 Vaccine + Activated T Cells
- After GI-4000 Vaccine #4 (Experimental): GI-4000 Monthly - For those with incomplete removal of tumor GI-4000 Monthly + Chemotherapy - For those with complete removal of tumor
  Interventions: Biological: Surgical Evaluation after Vaccine #4

INTERVENTIONS:
Other: Screening — A. SCREENING
  1. Consent
  2. Disease Evaluation (CT Scan/MRI; EGC/EUS; Laparoscopy)
  3. Physical Exam, History, Blood Tests
  4. Skin Test (for allergy to saccaromyces cerevisiae) yeast.
  5. Collection of Blood for research
  B. CHEMOTHERAPY AND RADIATION (as determined by Doctor)
  C. ENROLLMENT INTO ACTIVE PART OF STUDY
  1. Consent
  2. Chemotherapy
  3. GI-4000 Vaccine #1 + Prevnar + Activated T Cells
  4. GI-4000 Vaccine #2
  5. Disease Evaluation (CT Scan/MRI). If disease has spread, subject is taken off study. If disease is stable, subject go on to ARM A or ARM B.
  Arms: All Subjects
Biological: GI-4000 Vaccine — 1. Chemotherapy and Radiation
  2. GI-4000 Vaccine #3
  3. GI-4000 Vaccine #4
  Arms: ARM A
Biological: GI-4000 Vaccine + Activated T Cells — 1. Apheresis #2
  2. Chemoradiation
  3. Activated T Cells + GI-4000 Vaccine #3
  4. GI-4000 Vaccine #4
  Other Names: GI 4000 Vaccine; Activated T Cells
  Arms: ARM B
Biological: Surgical Evaluation after Vaccine #4 — SURGICAL EVALUATION (to determine disease status) A. For those who have complete removal of tumor. These subjects will continue to receive Chemotherapy AND GI-4000 Vaccination Monthly during Chemotherapy. Disease evaluation every 3-6 months (CT Scan/MR.
  B. For those sucjects who cannot have surgery or who have not had complete removal of tumor. These subjects will continue to have GI-4000 Vaccinations Monthly as long as there is no disease progression. Disease evaluation every 3-6 months (CT Scan/MR.
  Other Names: GI-4000 Vaccine
  Arms: After GI-4000 Vaccine #4

SUMMARY:
The purpose of this study is to determine if it is safe to add multiple immunotherapies to standard chemotherapy and radiation for treating pancreatic cancer tumors that cannot be completely removed by surgery.

1. GI-4000 Vaccination:

   The first involves a "vaccine," which is an injection (shot) that teaches your immune system to attack foreign invaders. The vaccine we will use is called "GI-4000" - a vaccine composed of yeast that is made to carry the same proteins (called "mutated Ras proteins") found in some pancreatic cancer cells.
2. Adoptive T-cell Transfer:

The second type of immunotherapy in this study is called "adoptive T-cell transfer." This involves collecting a specific type of white blood cells from you (called "T-cells")and growing T-cells grown in a lab which may help the research participants' immune systems recover more quickly after chemotherapy, and possibly improved response to other immunotherapies.

We hope that studying these agents together will teach us how to help the immune system fight pancreatic cancer.

DETAILED DESCRIPTION:
This Phase I/Pilot study will assess the safety and feasibility of the GI-4000 series vaccine with or without adoptive T cell transfer in subjects with locally advanced pancreatic cancer undergoing chemotherapy, radiotherapy, and surgical resection. Subjects will be randomized to either ARM A (GI-4000vaccine) or ARM B (GI-4000 vaccine and activated T cell transfer). All subjects will undergo apheresis of mononuclear cells immediately before receiving four cycles of gemcitabine/oxaliplatin (GemOx) chemotherapy ("immune preservation phase"). After the completion of chemotherapy, the apheresis product will be reinfused, and the subjects will enter the "priming phase," in which two biweekly doses (dose #1 and #2) of the appropriate GI-4000 vaccine (the one that best matches the mutations found in the patient's tumor) and a single dose of the Prevnar pneumococcal conjugate vaccine will be administered. At this time, those subjects who have not developed distant metastatic disease by CT/MRI will undergo chemoradiation, with ARM B subjects receiving a second apheresis immediately prior to the initiation of the chemoradiation. The pheresed product will be activated and expanded ex vivo and reinfused after chemoradiation is completed. All subjects will receive two more biweekly boosts of the GI-4000 vaccine (doses #3 and #4) while undergoing restaging with CT/MRI ("boosting phase"). Those who have not developed metastatic disease will undergo surgical evaluation for tumor resection. Patients who undergo R0 or R1 resection will receive up to three more weekly doses of GI-4000 prior to the initiation of adjuvant gemcitabine, monthly doses of GI-4000 during the four cycles of gemcitabine chemotherapy, and monthly GI-4000 doses thereafter. At the end of gemcitabine chemotherapy, apheresis will be performed for endpoint correlative studies. Those who are not candidates for surgery or whose tumors are not completely resected will continue to receive GI-4000 monthly booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with untreated, locally advanced pancreatic adenocarcinoma that expresses a GI-4000 related k-ras oncoprotein.

1. Histologically-confirmed pancreatic adenocarcinoma that expresses one of the GI-4000-related k-ras oncoproteins (G12V, G12C, G12D, Q61L, or Q61R)
2. Locally advanced disease, (stages I-III, i.e no evidence of metastasis outside the pancreas and its regional lymph nodes). Preferred subjects for entry into the study are those with borderline resectable disease, as defined by:

   * tumor that encases a short segment of the hepatic artery without extension to the celiac axis and that is amenable to resection and reconstruction, OR
   * tumor that abuts the superior mesenteric artery and that involves <180 degrees of the circumference of the artery, OR
   * short-segment occlusion of the superior mesenteric vein, portal vein, or their confluence with a suitable option available for vascular reconstruction because the veins are normal above and below the area of tumor involvement.
3. Age >18 years
4. ECOG performance status 0 or 1
5. Normal organ and bone marrow function as defined by:

   Absolute neutrophil count > 1,500/μl Platelets > 100,000/μl AST(SGOT)/ALT(SGPT)< 2.5 X institutional upper limit of normal Bilirubin < 2.0 mg/dL unless due to bile duct blockage by tumor Creatinine < 1.5 x ULN
6. A biliary stent 9F or biliary bypass before treatment, if tumor-related biliary obstruction is present
7. The ability to sustain adequate hydration and nutrition (>1500 cal/d) by oral intake or access for supplemental enteral feeding (nasoenteral tube, feeding jejunostomy or PEG)
8. Patients must have measurable disease by radiographic imaging, as defined by 1 lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20 mm with conventional techniques or 10 mm with spiral CT scanning. Marker elevation alone is insufficient for entry.
9. Ability to understand and the willingness to sign a written informed consent documents.
10. Adequate venous or catheter access and ability to tolerate apheresis.

Exclusion Criteria:

1. Tumor metastatic to peritoneum, liver or other organs
2. Tumor that is clearly resectable for curative intent
3. Prior chemotherapy, radiation therapy, targeted therapy, or immunotherapy for pancreatic cancer.
4. Receipt of any other investigational agents within 30 days prior to screening
5. Known HIV positive
6. A major surgical procedure or significant traumatic injury within 28 days prior to anticipated initiation of chemotherapy, an anticipated major surgical procedure during the course of the study, or a minor surgical procedure (laparoscopy, fine needle aspiration, or core biopsy) within 7 days of anticipated initiation of chemotherapy.
7. Serious non-healing wounds, ulcers, or bone fractures
8. Pregnancy or ongoing breast-feeding, as chemotherapy may pose substantial risk to the fetus/infant.
9. Patients whose treatment plan would require treating >50% of the liver to a dose greater than 30 Gy or treating > 50% of the total kidney volume to a dose greater than 18 Gy
10. Positive scratch test (immediate hypersensitivity, IgE mediated) to S. cerevisiae.
11. Active autoimmune disease requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of incorporating GI-4000 vaccine and activated T-cell infusion into a regimen of chemotherapy, radiation, and surgical resection to treat locally advanced pancreatic cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. O'Dwyer, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- See also: Abramson Cancer Center of the University of Pennsylvania — http://www.oncolink.com/